CLINICAL TRIAL: NCT05821166
Title: Moderate Whole-body Hyperthermia in Tumor Patients: Influence on Circulating Tumor Cells, Tumor Response, Quality of Life, Fatigue, Psyche, Immune Response and Tumor Microenvironment
Brief Title: Potential of Moderate Whole Body Hyperthermia to Enhance Response
Acronym: POWER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Sebastian Zschaeck, PD Dr. Sebastian Zschaeck, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POWER
Record Dates: First submitted 2023-02-07; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomization into intervention group (additional MWB-HT) and standard care (chemotherapy / immunotherapy) and control group (no MWB-HT), only standard care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mWBH (Experimental): patients receiving moderate Whole Body Hyperthermia
  Interventions: Device: moderate Whole Body Hyperthermia (mWBH)
- Control group (No Intervention): Patients do not receive moderate Whole Body Hyperthermia

INTERVENTIONS:
Device: moderate Whole Body Hyperthermia (mWBH) — Patients receiving 3-4 times mWBH
  Arms: mWBH

SUMMARY:
Using moderate whole-body hyperthermia (mWBH) in tumor patients to see the influence on circulating tumor cells, tumor response, quality of life, fatigue, psyche, immune response and tumor microenvironment

DETAILED DESCRIPTION:
Moderate whole-body hyperthermia (mWBH) is considered to be a very well-tolerated treatment. It has been used in numerous naturopathic and oncological practices for decades. It is also being used more and more with an increasing number of non-oncological diseases. A recently published randomized study was able to prove a sustained positive effect of whole-body hyperthermia in patients with depressive episodes. However, there are no clinical studies that demonstrate the benefit of this measure with regard to oncological treatment. There is also a lack of clarity about the mechanism of action of mWBH. A positive modification of the tumor microenvironment (increased perfusion, reduced interstitial pressure) and an increased activation of tumor-killing immune cells could be shown preclinically - however, a clinical evaluation of these mechanisms has not yet taken place.

This randomized study aims to evaluate the effect of mWBH on the tumor response of patients suffering from advanced cancer. The aim of the study is to demonstrate an improvement in the therapy response rate three months after the end of therapy through the additional use of mWBH, measured by a positive influence on the change in the number of circulating tumor cells from the time before therapy to the time three months after the start of therapy.

Quality of life reported by patients, recorded by the FACT-G questionnaire, as well as psychological parameters, fatigue and various other parameters with regard to an increase in the effect on the tumor are evaluated as secondary endpoints. All patients also receive serial immune monitoring. For this purpose, blood samples are taken before therapy and several times during the course of the therapy, which are then evaluated with regard to cytokines, immunological proteins and specific subgroups of immune cells.

The patients all receive guideline-based therapy in line with current internal practice. In addition to standard therapy, patients are randomized 1:1 and, if randomized to the mWBH arm, receive an additional 3-4 mWBH sessions during their oncological treatment. A total of six different patient groups are included, all with palliative therapy intentions (patients with multiple metastatic malignant melanoma before initiation of immunotherapy (checkpoint blockade), patients with metastatic or inoperable pancreatic carcinoma for whom first-line chemotherapy with FOLFIRINOX is planned, patients before palliative radiation therapy for a hormone-receptor-positive breast cancer who have previously received palliative systemic therapy and have at least one other tumor lesion in addition to the one that was irradiated, patients with metastatic sarcoma in whom ablation of the metastases is not possible and who are receiving palliative first-line therapy using Doxorubicin is planned to treat patients with metastatic or loco-regionally recurrent HPV-associated squamous cell carcinoma of the head and neck region, cervix, anus or vulva, for whom no local therapy methods are possible and palliative first-line platinum therapy is planned, patients with metastatic castration-resistant prostate cancer with progressive disease after exhaustion of recommended therapy options for whom a therapeutic trial with lutetium-177-PSMA has been indicated). A total of at least 72 patients, stratified into the 6 subgroups mentioned above, should be evaluated in the study, who should receive three to four sessions of mWBH in addition to standard oncological treatment. In order to obtain the necessary minimum number of patients in all subgroups, the inclusion of 80 patients in the study is necessary with an expected drop-out rate of 10%.

In order to record the effect of mWBH on quality of life, fatigue and depression, study participants must fill out a questionnaire on quality of life, fatigue and depression before the start of therapy, at the end of treatment and two weeks after therapy. To evaluate the influence of mWBH on immune parameters, patients also receive additional blood samples before the start of therapy, at the end of therapy and at two follow-up times, which can normally be combined with routine blood samples.

For further risk stratification, the samples obtained after an operation or biopsy can be used for further analysis. This examination means no additional intervention and no increased risk for the patient, since these have already been carried out routinely. Patients have the option of expressly agreeing to the removal and further use of these biomarkers or rejecting them as part of the declaration of consent.

ELIGIBILITY:
Inclusion Criteria:

* The general condition of the patients must be sufficient for multimodal treatment (corresponding to WHO status 0-2)
* Tumordisease in a palliative setting of the following 6 groups:

  1. Malignant melanoma, treatment-naive stage IV with multiple metastases and missing BRAF-V600 mutation. With indication for initiation of immunotherapy using PD-1 and CTLA-4 antibody therapy.
  2. Patients with metastatic or inoperable pancreatic cancer, who are planning first-line chemotherapy with FOLFIRINOX is.
  3. Patients with an indication for palliative radiation therapy extracranial, tumor manifestation with a prescribed radiation dose of 30 to 36 Gy due to hormone receptor-positive carcinoma of the breast, patients must have at least one additional (marker) lesion not treated with radiation.
  4. Patients with metastatic high-grade sarcoma for whom metastasis-directed ablative therapy methods are not possible and palliative first-line therapy with doxorubicin.
  5. Patients with metastatic or loco-regionally recurrent HPV-associated squamous cell carcinoma (of the head and neck region, cervix, anus or vulva) for whom local therapies are not possible and for whom palliative first-line therapy containing platinum is planned.
  6. Patients with metastatic, castration-resistant prostate cancer, with progressive disease after exceeding the recommended therapy options for which a therapy attempt with lutetium-177-PSMA was indicated.

Exclusion Criteria:

* Presence of contraindications to simultaneous chemotherapy or whole-body hyperthermia
* Serious or active comorbidities that could interfere with treatment or understanding of the nature and content of the study, for example:

  * Chronic inflammatory bowel disease
  * Acute infections
  * Serious cardiovascular or pulmonary comorbidities
  * Mental illnesses, showing the proper Study participation or recording the nature of the study to make impossible
  * Presence of cerebral metastasis
  * Diabetes mellitus with risk of end-organ damage

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
change in the number of circulating tumor cells before therapy vs after therapy | Test therapy naive versus three months after the start of therapy
  ANCOVA is used as the statistical methodology. The change in the number of circulating tumor cells three months after the start of therapy is the dependent variable, the group (intervention or control) and the number of circulating tumor cells as well as the tumor entity (6 groups) are independent variables. Case number estimation: So far there are no studies that have examined this outcome. We assume that the intervention effect is moderate and that an effect size of 0.6 to 0.7 can be achieved.
  If 36 patients per arm are included in the study, an effect size (Cohen's d) of 0.67 or greater at a two-sided significance level of α=0.05 with a power of 80% can be demonstrated using the t-test for independent samples.

SECONDARY OUTCOMES:
Response of the tumors | three months after the start of therapy
  morphologically in imaging
Quality of life of the patients | measured before and 2 weeks after the end of therapy (end of therapy is determined as the last planned mWBH session) or at a comparable time in the control group
  The hypothesis is that patients with mWBH report a higher quality of life than patients without mWBH. Life Quality will be assessed in a standardized questionnaire as EORTC QLQ-30
influence of mWBH on depressive/dysthymic moods/episodes as well as on fatigue symptoms | Follow-up visits, in total 2 years follow up time
  reported by patients in standardized questionnaire
impact of patient-reported organ-specific functional impairment | Follow-up visits, in total 2 years follow up time
  measured by standardized questionnaires (depending tumor entity e.g. PR25 in patients with prostate cancer, BR23 in breast cancer, MEL38 in melanoma, and PAN26 in pancreatic cancer
influence of mWBH on different leukocyte sub-populations and the plasma concentration of cytokines/proteins, which indicate a suspected predictive effect on the response to immunotherapy. | measurement before treatment compared with the one after treatment
  leukocyte sub-populations are measured by FACS
side effect profile of mWBH | during and after treatment in Follow-up visits, in total 2 years follow up time
  side effects reported by practitioner and the patient, potential side effects will be documented in Case Report Form (CRF) which will be filled out in follow up visits
Tumor marker responses in patients who have measurable tumor markers that have previously also been correlated with disease activity | measurement before treatment compared with the one after treatment
  It is assumed that this is the case in a total of 50 patients (ITT) (25 in each group)
survival rate and rate of progression-free surviving patients across all stratification groups. | 1 and 2-year
  PFS = death or any form of tumor recurrence, local or systemic, are counted as an event here
The impact of mWBH on leukocyte nadir and time to recovery in patients receiving radiation, lutetium, or cytostatic therapy (arms 2-6) | during and after treatment in blood assessment
  Comparison of routine lab-testing within intervention group and between control
In arm 3 (breast cancer): The influence of mWBH on the occurrence of an abscopal effect, i.e. a response of a tumor lesion outside the irradiated volume (dose < 4 Gray during fractionated palliative irradiation) | in follow-up routine imaging controls ( e.g. 3 months after treatment)
  Response is evaluated by the RECIST criteria: CR or PR

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik für Radioonkologie und Strahlentherapie, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No